CLINICAL TRIAL: NCT05396235
Title: A Clinical Pharmacology Study of MT-3921 in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MT-3921-Z-101; jRCT2031220182 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2022-05-22; First posted 2022-05-31 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Healthy Adult Males

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT-3921 (Experimental): Intravenous (IV)
  Interventions: Biological: MT-3921
- Placebo (Placebo Comparator): Intravenous (IV)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MT-3921 — Solution for infusion; Intravenous (IV)
  Other Names: Unasnemab
  Arms: MT-3921
Biological: Placebo — Solution for infusion; Intravenous (IV)
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and pharmacokinetics when MT-3921 or a placebo is intravenously given to Japanese healthy adult male subjects

ELIGIBILITY:
Inclusion Criteria: Additional screening criteria check may apply for qualification:

* Japanese healthy adult males
* Subjects aged between 18 and 55 years inclusive at the time of informed consent
* Subjects with a full understanding of the nature of this study who have consented in writing to participate in the study

Exclusion Criteria: Additional screening criteria check may apply for qualification:

* Subjects with or having a history or treatment history of disorders, including cardiac, hepatic, renal, gastrointestinal, respiratory, neuropsychiatric, hematopoietic, or endocrine system disorder, who are judged by the investigator (or subinvestigator) to be unfit for study participation
* Subjects with a history of drug or food allergies, including anaphylaxis or significant allergic reactions
* Subjects with a body mass index (BMI) of less than 18.5 kg/m^2 or greater than 25 kg/m^2 at the time of screening or Day -1 or those with a body weight of less than 50 kg or greater than 80 kg
* Subjects who have donated blood or from whom blood samples have been collected in a total amount of 400 mL or more within 12 weeks prior to informed consent, 200 mL or more within 4 weeks prior to informed consent, or 800 mL or more within 1 year prior to informed consent
* Subjects who have donated blood component or platelet apheresis within 2 weeks prior to informed consent
* Subjects with or having a history of drug dependence or alcohol dependence
* Subjects with clinically significant abnormalities on a 12-lead ECG, with a Fridericia-corrected QT (QTcF) interval of ≥450 msec, or with clinically significant abnormalities on an auscultation
* Subjects with a positive result for hepatitis B virus surface (HBs) antigen, serological test for syphilis, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen/antibody at screening
* Subjects with a positive polymerase chain reaction (PCR) test for Coronavirus disease 2019 (COVID-19)
* Subjects with a family history of sudden death
* Subjects who answered "yes" to any of the items of suicide ideation or suicide attempts in the Columbia Suicide Rating Scale (C-SSRS) assessment in the screening period
* Subjects who do not agree to practice contraception during the study period
* Subjects who have previously received anti-RGMa antibodies, including this investigational product
* Subjects who have participated in other clinical studies and received other investigational products within 12 weeks before informed consent
* Subjects who have used any drug other than the investigational product in the period within 7 days before the start of investigational product administration or 5 times the half-life of the drug, whichever is longer

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2022-12-24 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with adverse events | 16 weeks
Percentage of subjects with adverse reactions | 16 weeks
Time course of serum concentrations of MT-3921 | Day 1, 2, 3, 4, 8, 15, 29, 57, 85, and 113.

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No